CLINICAL TRIAL: NCT06894394
Title: Implementing a Group Version of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) in a Spanish Day Hospital for Adolescents With Severe Mental Disorders.
Brief Title: Group Version of the UP-A in a Spanish Day Hospital for Adolescents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Julia García Escalera, Professor, Universidad Nacional de Educación a Distancia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-PSI-2023/2
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Disorders; Depressive Disorder; Emotional Disorder
Keywords: Unified Protocol; Emotional Disorders; Adolescents; Severe mental disorders; Day Hospital; UP-A; Spain
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Intervention Group of an uncontrolled study.
  Interventions: Behavioral: UP-A

INTERVENTIONS:
Behavioral: UP-A — The UP-A (Ehrenreich-May et al., 2018, 2020, 2022) is a transdiagnostic intervention with eight modules targeting neuroticism. It improves emotion regulation and reduces avoidance, with summaries after each module and a Parent Module (P). The intervention is a group adaptation of the Spanish version of UP-A that consists of 16 weekly sessions, each lasting 60 to 90 minutes, held in person at a Day Hospital within the Spanish public healthcare system. Due to the complexity of the setting, parent sessions are not viable. However, parents receive summaries of the modules covered with the adolescents, as well as the Parent Module (Parenting the Emotional Adolescent), to support their understanding of the treatment content.

SUMMARY:
This study aims to adapt the Spanish version of the UP-A for group delivery in an intensive treatment setting for adolescents with severe mental disorders within a day hospital of the Spanish public healthcare system. It also explores the feasibility and clinical utility of this adaptation through an uncontrolled study with pre-post and follow-up assessments (at 3, 6 and 12 months). The evaluation includes anxiety, depression, transdiagnostic variables, engagement, and satisfaction from adolescents, parents, and clinicians, as well as changes in adolescents' primary problems.

DETAILED DESCRIPTION:
Anxiety and depression are among the most prevalent mental health disorders in adolescents, often co-occurring due to shared transdiagnostic factors such as poor emotion regulation, high negative affect, and cognitive avoidance. When severe, these disorders significantly increase the risk of self-harm and suicide, which is a leading cause of death among young people worldwide. Given these risks, it is crucial to develop interventions that effectively target these transdiagnostic mechanisms and improve access to treatment for adolescents with severe emotional disorders.

The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) was designed to target neuroticism, a key vulnerability factor in emotional disorders. While the UP-A was originally developed as an individual treatment, its adaptation to a group format could enhance accessibility and optimize mental health resources. Although the UP has been successfully implemented in group settings for adults, there is limited research on the feasibility of a group-based UP-A intervention, particularly in clinical settings with adolescents experiencing severe mental health conditions.

This study aims to adapt the Spanish version of the UP-A to a group format in an intensive treatment setting, specifically within a day hospital of the Spanish public healthcare system, where adolescents receive comprehensive, multidisciplinary care for severe emotional disorders. The study also explores the feasibility and clinical utility of this adaptation through an uncontrolled study, assessing pre-post and follow-up outcomes in two consecutive groups. The intervention consists of 16 weekly sessions, each lasting 60 to 90 minutes.

The study evaluates changes in anxiety, depression, transdiagnostic variables (e.g., emotional avoidance, emotion regulation strategies), engagement, and satisfaction from the perspectives of adolescents, parents, and clinicians. Additionally, adolescents' self-rated primary problems and clinicians' assessments of overall clinical progress were analyzed. Follow-up assessments will be conducted 3, 6 and 12 months post-intervention to measure sustained effects.

ELIGIBILITY:
Inclusion Criteria:

* Being an active patient at the Day Hospital of the Puerta de Hierro Hospital
* Presenting, as the main diagnosis (most serious diagnosis or the one that interferes the most), an emotional disorder with moderate or high severity including the following disorders based on DSM-5 categories: Depressive Disorders (Major Depressive Disorder and Persistent Depressive Disorder), Bipolar Disorders (Bipolar I and II Disorder, Cyclothymic Disorder), Anxiety Disorders (Specific Phobia, Panic Disorder, Agoraphobia, Social Anxiety Disorder, Generalized Anxiety Disorder), Obsessive-Compulsive and Related Disorders (including Body Dysmorphic Disorder, Hoarding Disorder, Trichotillomania and Excoriation (Skin-Picking) Disorder), Trauma and Stressor-Related Disorders (Reactive Attachment Disorder, Post-Traumatic Stress Disorder, Acute Stress Disorder and Adjustment Disorders), Dissociative Disorders (Dissociative Identity Disorder, Depersonalization/Derealization Disorder) and Somatic Symptom and Related Disorders (Somatic Symptom Disorder and Illness Anxiety Disorder). Specified and unspecified disorders from the above categories are also included.
* Being able to participate normally in group therapy (despite presenting self-harm or suicidal ideation, severe depressive disorder or dysfunctional personality and/or autism spectrum disorder)
* Being 11-18 years of age
* Being proficient in Spanish
* Being able to attend the evaluation and treatment sessions
* At least one of the adolescent's parents or legal guardians being able to complete the evaluation questionnaires
* If the participant was taking psychiatric medication, the dose being remaining stable for at least 1 month before the start of treatment and throughout it

Exclusion Criteria:

* Presenting one or more of the following clinical conditions (either as a main or comorbid diagnosis): 1) Intellectual Disability, 2) Autism Spectrum Disorder accompanied by an intellectual disability that does not allow for group therapeutic work, 3) Disruptive, Impulse-Control and Conduct Disorders with a severity level that hinders group work, 4) Eating Disorders as the main diagnosis, 5) Psychotic Spectrum Disorders or psychotic-type symptoms, 6) Substance Abuse Disorders (excluding cannabis, coffee and/or nicotine) as the main diagnosis
* The characteristics or severity of the symptoms presented by the adolescent requiring an individual intervention or one adapted to the specific clinical condition
* Suffering from a serious medical illness that makes the adolescent's participation in the treatment program unsustainable
* The participant, or, if under 16 years of age, his or her parents, having refused to sign the informed consent

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in Anxiety and Depressive Symptoms as Assessed by RCADS-30 | Up to 12 months
  The Revised Child Anxiety and Depression Scale-30 (RCADS-30; Sandín et al., 2010) at pre, post-intervention and 3, 6 and 12 months follow-up.
  Range from 0 to 90. Symptoms of anxiety (panic disorder, social phobia, separation anxiety disorder, generalized anxiety disorder, and obsessive-compulsive disorder) and depressive disorders symptoms. Higher scores mean a worse outcome.
  Parents completed the "parent version" of the RCADS.
Changes in Anxiety and Depressive Symptoms's Interference as Assessed by EIDAN | Up to 12 months
  Depression and Anxiety Interference Scale for Children and Adolescents EIDAN (Espinosa et al., 2022) . It is a 10-item self-reported instrument that evaluates the interference of emotional symptoms in the adolescent's daily functioning in the previous weeks, in several contexts (school, family and with peers). The higher the score, the higher the level of interference. Assessed at pre, post-intervention and 3, 6 and 12 months follow-up.
  Range from 10 to 40. Parents completed the "parent version" of the EIDAN.
Top Problems Measure | Up to 12 months
  The adolescent version of the Top Problem Assessment (TPA) (Ehrenreich, 2018; adapted from Weisz et al., 2011) was used to enhance treatment outcomes and strengthen the therapeutic alliance. Adolescents were asked to write down the issues that concerned them the most and assess the severity of each problem by rating its impact on daily functioning on a scale from 0 ("not a problem at all") to 10 ("very, very much a problem"). Each adolescent selected between one and three problems and evaluated their severity at five time points: at the beginning of the program (session 3), mid-treatment (session 8), the final session (session 16), and during follow-ups at 3, 6 and 12 months.
Changes in Emotion Regulation Strategies as Assessed by CERE | Up to 12 months
  Emotion Regulation Strategies Questionnaire CERE-II (Sandín et al., 2008). Adapted to Spanish by Sandín et al. (2008).
  Evaluates 7 subscales of the "emotion regulation" construct at pre, post-intervention and 3, 6 and 12 months follow-up.
  Higher scores in maladaptive regulation strategies (supression; rumination; distraction) and lower scores in adaptive strategies (attention/awareness/understanding; acceptance/tolerance; cognitive reappraisal; self-instructions) mean a worst outcome

SECONDARY OUTCOMES:
Changes in Positive and Negative Affect as Assessed by PANASN | Up to 12 months
  he Children Positive and Negative Affect Schedule [Escalas PANAS para niños y adolescentes] (PANASN; Sandín, 2003) at pre, post-intervention and 3, 6 and 12 months follow-up. Positive and negative affect.
  Range 10-30. Higher scores of negative affect and lower scores os positive affect mean a worse outcome.
Changes in Depressive Symptoms as Assessed by CDN | Up to 12 months
  The Depression Questionnaire for Children and Adolescents [Cuestionario de Depresión para Niños y Adolescentes] (CDN; Sandín et al., 2016) at pre, post-intervention and 3, 6 and 12 months follow-up.
  Depressive symptoms. Range from 0 to 48. Higher scores mean a worse outcome
Changes in Anxiety Sensitivity as Assessed by CASI | Up to 12 months
  Childhood Anxiety Sensitivity Index CASI (Silverman et al., 1991) ; Spanish adaptation by (Sandín et al., 2002). Anxiety sensitivity at pre, post-intervention and 3, 6 and 12 months follow-up.
  Range 18 to 54. Higher scores mean a worse outcome.
Changes in Emotional Avoidance as Assessed by EASI | Up to 12 months
  Emotional Avoidance Strategy Inventory for Adolescents EASI-A ( Kennedy & Ehrenreich-May, 2017) ; Spanish adaptation by (García-Escalera et al., 2016). Emotional avoidance strategies at pre, post-intervention and 3, 6 and 12 months follow-up.
  Range 0 to 68. Higher scores mean a worse outcome.
Changes in Satisfaction with Life as Assessed by SWLS | Up to 12 months
  Satisfaction with Life Scale SWLS (Diener et al., 2010; adapted to Spanish by Sandín et al., 2015).
  Evaluates satisfaction with life at pre, post-intervention and 3, 6 and 12 months follow-up. Range 5 to 20. Lower scores mean a worse outcome.
Changes in Attachment Styles as Assessed by ARSQ | Up to 12 months
  Adolescent Relationships Scales Questionnaire ARSQ (Scharfe, 1999) ; adapted to Spanish by (Magaz et al., 2011). The ARSQ is an instrument composed of 17 self-reported items, which allows obtaining scores for the three types of attachment identified in the theory of Bartholomew (1990) and Bartholomew and Horowitz (1991): secure attachment, fearful/preoccupied attachment, and avoidant attachment. Evaluates attachment styles at pre, post-intervention and 3, 6 and 12 months follow-up.
  Higher scores in insecure attachment styles (fearful/preoccupied attachment, and avoidant attachment) and lower scores in secure attachment style mean a worst outcome.
Changes in Somatic Symptoms as Assessed by PHQ-15 | Up to 12 months
  Somatic Symptoms Scale extracted from the PHQ-15, Patient Health Questionnaire (adapted from the patient health questionnaire - physical symptoms - PHQ-15; (Kroenke et al., 2002) ; Extracted and translated from the APA website - DSM-5 Level 2 Cross -Cutting Symptom Measures). It is composed of 13 items that evaluate somatic symptoms in adolescents between 11 and 17 years old at pre, post-intervention and 3, 6 and 12 months follow-up. Range 0 to 26. Higher scores mean a worse outcome.
Changes in Severity of Clinical Diagnosis as Assessed by CSR | 16 weeks
  The Clinician Severity Rating CSR (ADIS-IV Interview; Silverman et al., 2008). This scale indicates, for each main and secondary diagnosis, the clinician's estimate of severity according to the following scale from 0 to 8: 0 = no seriousness, 1 - 2 = little disturbance/no disabling, 3 - 5 = clear disturbance/disabling (at least a 4 is required for diagnosis) 6 - 7 = high/disabling disturbance; 8 = very serious/disabling disturbance.
  Assessed at pre and post-treatment.
Changes in Level of Functioning as Assessed by CGAS | Up to 12 months
  The Children's Global Assessment Scale CGAS (Schaffer et al., 1983; version translated into Spanish by the Xunta de Galicia Agreement and the University of A Coruña Foundation, 2012). It is a clinician-estimated measure of the adolescent's overall level of functioning in the last month. Scores range from 100-91 (optimal functioning in all areas) to 10-1 (constant need for supervision).
  Evaluates General Functioning at pre, post-intervention and 3, 6 and 12 months follow-up.
Changes in Clinician Estimated Severity of Anxiety and Depressive Symptoms as Assessed by CGI-S | Up to 12 months
  The Clinical Global Impression (Severity) Scale CGI-S (Guy, 1976) . Using this scale, the clinician estimated the severity of the adolescent's anxiety and depression symptoms. Scores will range from 1 ("Normal, not at all ill"), to 7 ("Extremely ill").
  Evaluated at pre, post-intervention and 3, 6 and 12 months follow-up.
Changes in Clinician Estimated Improvement of Anxiety and Depressive Symptoms as Assessed by CGI-I | Up to 12 months
  The Clinical Global Impressions (Improvement) Scale CGI-I (Guy, 1976) . This scale was completed by the clinicians during post-treatment and follow-ups. The adolescent's improvement was scored on a scale from 1 to 7, with 1 being "very much improved" and 7 being "very much worse".
  Assessed at post-intervention and 3, 6 and 12 months follow-up.
Satisfaction with the program and therapeutic alliance | 16 weeks
  In the post-treatment evaluation, adolescents and involved parents completed a 12-item questionnaire that evaluates satisfaction with the program and the quality of the relationship with the therapist (Sandín et al., 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M. Valiente, Professor, Study Director — Universidad Nacional de Educación a Distancia
Locations (1):
- Hospital de Día Infantojuvenil del Hospital Puerta de Hierro de Majadahonda, Madrid, Madrid, Spain